CLINICAL TRIAL: NCT06674317
Title: Tailoring an Internet Delivered Cognitive Behavioral Therapy for Insomnia in Persons with Inflammatory Rheumatic Diseases: Acceptability and Feasibility- Phase 2
Brief Title: Tailoring an Internet Delivered Cognitive Behavioral Therapy for Insomnia in Persons with Inflammatory Rheumatic Diseases
Acronym: REPOSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Deborah Da Costa, Deborah Da Costa, PhD, Associate Professor, Department of Medicine, McGill University; Scientist, RI-MUHC, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-6547
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Group 1: I-CBTi group: This group you will have access to the internet delivered cognitive behavioral therapy for insomnia intervention following the completion of the first study entry questionnaire.
  Group 2: WLC group: This group will be offered access to the internet delivered cognitive behavioral therapy for insomnia intervention AFTER completion of the third online questionnaires 5 months after group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Internet delivered Cognitive Behaviour Therapy for Insomnia group (Experimental): This group you will have access to the internet delivered cognitive behavioral therapy for insomnia intervention following the completion of the first study entry questionnaire.
  Interventions: Behavioral: Internet Delivered Cognitive Behavioral Therapy for Insomnia in Persons with Inflammatory Rheumatic Diseass
- Arm 2: Wait list Control Group (Other): This wait list control group will be offered access to the internet delivered cognitive behavioral therapy for insomnia intervention AFTER completion of the third online questionnaires 5 months after group assignment.
  Interventions: Behavioral: Internet Delivered Cognitive Behavioral Therapy for Insomnia in Persons with Inflammatory Rheumatic Diseass

INTERVENTIONS:
Behavioral: Internet Delivered Cognitive Behavioral Therapy for Insomnia in Persons with Inflammatory Rheumatic Diseass — Cognitive behavioral therapy for insomnia (CBTi) is considered a first-line treatment for insomnia. Access to this treatment option is limited therefore we have been developing an internet delivered cognitive behavioral therapy for insomnia (I-CBTi) to help overcome accessibility barriers.
  The purpose of this study is to pilot test a tailored internet-delivered cognitive behavioral therapy for insomnia (I-CBTi) intervention for persons with Inflammatory Rheumatic Diseases showing symptoms of insomnia.

SUMMARY:
Cognitive behavioral therapy for insomnia (CBTi) is considered a first-line treatment for insomnia. Access to this treatment option is limited therefore the investigators have been developing an internet delivered cognitive behavioral therapy for insomnia (I-CBTi) to help overcome accessibility barriers.

The purpose of this study is to pilot test a tailored internet-delivered cognitive behavioral therapy for insomnia (I-CBTi) intervention for persons with Inflammatory Rheumatic Diseases showing symptoms of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported physician diagnosis of one or more of the following Inflammatory Rheumatic Diseases: rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis or other spondyloarthropathies, systemic lupus erythematosus
* Have an e-mail address and internet access
* Speak and read English or French
* Resident of Canada and living in Canada for the duration of the trial
* Have insomnia symptoms ( score ≥8 on the Insomnia Severity Index (ISI) )

Exclusion Criteria:

* Self-reported sleep disorder diagnosed by a physician other than insomnia (e.g. obstructive sleep apnea)
* Severe psychiatric disorder (e.g. schizophrenia, bipolar disorder) or neurological disorders (e.g diagnosis of dementia, Parkinson disease, epilepsy)
* Already involved in psychotherapy addressing sleep difficulties
* Shift work in the past 3 months or next 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Participant Acceptability of the Internet Delivered Cognitive Behavioral Therapy for Insomnia (CBTi) Intervention as Assessed by the Treatment Expectancies and Perceived Credibility Questionnaire (TEPCQ) | At enrollment
  The Treatment Expectancies and Perceived Credibility Questionnaire (TEPCQ) is a 5-item questionnaire that evaluates participants' therapeutic expectancies and the credibility they give to the treatment proposed.
Participant Acceptability of the Internet Delivered Cognitive Behavioral Therapy for Insomnia (CBTi) Intervention as Assessed by the Treatment Perception Questionnaire (TPQ) | From enrollment until 8 weeks post treatment
  The Treatment Perception Questionnaire (TPQ) assesses the degree to which participants consulted the written and visual content of each module in the internet delivered Cognitive Behavioral Therapy for Insomnia program, the usefulness of each of the 6 modules, level of satisfaction with the written and video content, as well as the global satisfaction with the intervention.
Change in Sleep Difficulty from Enrollment to 3 Months Post Treatment as Assessed by the Sleep Severity Index (ISI) | Enrollement to 3 months post treatment
  The Insomnia Sleep Index is a 7-item self-report questionnaire measuring the perceived severity and difficulties with sleep. The measure yields a total score from 0-28. Scores from 0-7 indicate no insomnia, 8-14 subthreshold insomnia, 15-21 moderate clinical insomnia and 22-28 severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Da Costa, PhD, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: No